CLINICAL TRIAL: NCT00639418
Title: An Observational Study to Describe Pediatric Influenza Vaccine Coverage Among Pediatricians in the United States
Brief Title: A Study to Describe Pediatric Influenza Vaccine Coverage
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MI-MA156
Record Dates: First submitted 2008-03-04; First posted 2008-03-20 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Participants 6 to 23 months: Pediatric influenza vaccine coverage within practicing pediatricians' offices for participants 6 to 23 months of age
  Interventions: Biological: Influenza vaccination
- Participants 24 to 59 months: Pediatric influenza vaccine coverage within practicing pediatricians' offices for participants 24 to 59 months of age
  Interventions: Biological: Influenza vaccination
- Participants 5 to 8 years: Pediatric influenza vaccine coverage within practicing pediatricians' offices for participants 5 to 8 years of age
  Interventions: Biological: Influenza vaccination
- Participants 9 to 17 years: Pediatric influenza vaccine coverage within practicing pediatricians' offices for participants 9 to 17 years of age
  Interventions: Biological: Influenza vaccination

INTERVENTIONS:
Biological: Influenza vaccination — This non-interventional study prospectively captured vaccine coverage and practices of participating physician offices through use of surveys during the influenza vaccination season.

SUMMARY:
The purpose of this study is to describe flu vaccine coverage in children under 18 years of age and to examine correlations between in-office flu vaccine coverage and the use of various tactics to increase vaccine coverage.

DETAILED DESCRIPTION:
To describe influenza vaccine coverage in children less than 18 years of age in practicing pediatricians' offices and family medicine physicians' offices and to examine correlations between in-office influenza vaccine coverage and the use of various tactics to increase vaccine coverage.

ELIGIBILITY:
Sites selected to participate were required to be able to accurately identify the number of patients under their care by age group and provide influenza vaccine at their location.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physician offices that were selected to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 147494 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Ambrose, M.D., Study Director — MedImmune LLC
Locations (187):
- United States (187):
  - Ark-La-Tex Pediatric Research, Birmingham, Alabama
  - Jordan Ridge Kids and Teens, Daphne, Alabama
  - Pediatrics by the Bay, Daphne, Alabama
  - Montgomery Pediatric Associates, PA, Montgomery, Alabama
  - Tennessee Valley Pediatric Associates, Sheffield, Alabama
  - Carlile Pediatrics, Wetumpka, Alabama
  - Adventures in Pediatrics, Wasilla, Alaska
  - Pendleton Pediatrics, Chandler, Arizona
  - Armadillo Pediatrics, Phoenix, Arizona
  - Grayhawk Pediatrics, Scottsdale, Arizona
  - North Scottsdale Pediatrics Associates, Scottsdale, Arizona
  - Papago Buttes Pediatric Center PC, Scottsdale, Arizona
  - Cholla Pediatrics, Tucson, Arizona
  - Central Arkansas Pediatric Clinic, Benton, Arkansas
  - Bentonville Pediatrics, Bentonville, Arkansas
  - Children's Investigational Research Program, Bentonville, Arkansas
  - The Pediatric Clinic, North Little Rock, Arkansas
  - Adventures in Pediatrics, Wasilla, Arkansas
  - Gardens Medical Center, Bell Gardens, California
  - Pratima Patel, MD, Covina, California
  - Mission Care Pediatrics, Folsom, California
  - Razia Sheikh, Fresno, California
  - Del Rosario Medical Clinic, Inc., Huntington Park, California
  - Ching Ti, M.D., Oceanside, California
  - Providence Pediatrics, Poway, California
  - Stonestown Pediatrics, San Francisco, California
  - Eugene I Litwer, Santa Ana, California
  - Louella Peckson, MD, Van Nuys, California
  - Pediatric Partners of the Southwest, Durango, Colorado
  - Evergreen Pediatrics, Evergreen, Colorado
  - Children's Clinic of Pueblo, Pueblo, Colorado
  - Darien Pediatric Associates, Darien, Connecticut
  - Norwich Pediatric Group PC, Norwich, Connecticut
  - Prospect Family Practice, Prospect, Connecticut
  - Bay Street Pediatrics, Westport, Connecticut
  - JFK Pediatrics, Atlantis, Florida
  - Giangreco, Scarano & Taylor Pediatrics, Bradenton, Florida
  - Kids and More Pediatric Care, Brandon, Florida
  - Sawgrass Pediatrics, Coral Springs, Florida
  - Ramon Maldonado, MD, Homestead, Florida
  - Atlantic Coast Pediatrics, Merrit Island, Florida
  - Guillermo S. Llosa, MD PA, Miami, Florida
  - The Pediatric Specialists Medical Group, New Port Richey, Florida
  - Orange Park Pediatrics, Orange Park, Florida
  - Childrens Medical Association, Plantation, Florida
  - St Pete Pediatrics, St. Pete Beach, Florida
  - Lynne Ellis, St. Petersburg, Florida
  - Wesley Chapel Internal Medicine & Pediatrics PA, Wesley Chapel, Florida
  - KidCare Pediatrics, LLC, College Park, Georgia
  - Jesup Pediatrics, Jesup, Georgia
  - Pediatric and Adolescent Healthcare, PC, Marietta, Georgia
  - Sandy Plains Pediatrics, Ringgold, Georgia
  - Zaman Pediatric Center, Snellville, Georgia
  - DuPage Pediatrics, Darien, Illinois
  - Alzein Pediatrics, Evergreen Park, Illinois
  - Mary E. Lewis MD. PC, LaGrange, Illinois
  - Lake Shore Pediatrics, Libertyville, Illinois
  - Port City Pediatrics, Muskegon, Illinois
  - North Suburban Family Healthcare, Vernon Hills, Illinois
  - Pediatric Associates Inc, Fort Wayne, Indiana
  - Northpoint Pediatrics, Indianapolis, Indiana
  - Jeffersonville Pediatrics, Jeffersonville, Indiana
  - Del Pilar Medical & Urgent Care Center, Mishawaka, Indiana
  - RMH Pediatrics, Rushville, Indiana
  - MercyCare Edgewood, Cedar Rapids, Iowa
  - Alegent Health Clinic, Council Bluffs, Iowa
  - St. John's Pediatrics, Leavenworth, Kansas
  - Paul J. Janson, MD, Florence, Kentucky
  - Oldham County Pediatrics, La Grange, Kentucky
  - Associates in Pediatrics, Baton Rouge, Louisiana
  - Ark-La-Tex Pediatric Research, Bossier City, Louisiana
  - Family Practice Pediatric Clinic, Lake Providence, Louisiana
  - Allstar Pediatrics (LEESVILLE, LA), Leesville, Louisiana
  - Pearl Acres Pediatrics, Slidell, Louisiana
  - Mecosta Health Services, Big Rapids, Michigan
  - Deckerville Health Services, Deckerville, Michigan
  - Port City Pediatrics, Muskegon, Michigan
  - Merrillwood Pediatrics, Royal Oak, Michigan
  - Northern Lights Pediatrics, Vadnais Heights, Minnesota
  - Tots Thru Teens, Bridgeton, Missouri
  - Priority Care Pediatrics, Kansas City, Missouri
  - Preferred Pediatrics, Lee's Summit, Missouri
  - Country Corner Family Medical Center, Mount Vernon, Missouri
  - Midwest Allergy and Asthma Clinic, Omaha, Nebraska
  - Henderson Pediatrics, Henderson, Nevada
  - Anthem Pediatrics, Henderson, Nevada
  - Harold Naiman, MD, Las Vegas, Nevada
  - Mediterranean Pediatrics, East Orange, New Jersey
  - Ronald M. Frank, MD, PA, Green Brook, New Jersey
  - Plaza Pediatrics, North Brunswick, New Jersey
  - New Beginnings Pediatrics, Phillipsburg, New Jersey
  - Pediatric Associates of New Jersey, Vineland, New Jersey
  - Four Seasons Pediatrics, Clifton Park, New York
  - Delmar Family Medicine, Delmar, New York
  - Prime Care Physicians, Delmar, New York
  - Perinton Pediatrics, Fairport, New York
  - Park Pediatrics, Floral Park, New York
  - Garden City Pediatric, Garden City, New York
  - ProKids, LLP, Levittown, New York
  - Clarkstown Pediatrics, New City, New York
  - North Court Pediatrics, North Syracuse, New York
  - Orchard Park Pediatrics, Orchard Park, New York
  - Pomona Pediatrics, Pomona, New York
  - Edward Lewis, M.D., P.C., Rochester, New York
  - Asheboro Research Associates, Asheboro, North Carolina
  - Asheville Pediatric Association, Asheville, North Carolina
  - Blue Ridge Pediatric and Adolescent Medicine, Beone, North Carolina
  - Cornerstone Medical Center, Burlington, North Carolina
  - Cary Medical Research, Cary, North Carolina
  - Haywood Pediatrics, Clyde, North Carolina
  - Lucas Pediatrics, Greensboro, North Carolina
  - Briargate Medical Associates, Greensboro, North Carolina
  - Northwest Pediatrics, Inc., Greensboro, North Carolina
  - Rainbow Pediatrics, Henderson, North Carolina
  - Blue Ridge Community Health Services, Hendersonville, North Carolina
  - Mountain View Pediatrics, P.A., Morganton, North Carolina
  - Masoud Ahdieh MD, Rockingham, North Carolina
  - Columbus Pediatrics and Adolescent Care, Whiteville, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Kids First Pediatrics, Canfield, Ohio
  - Shipley Child Health Clinic, Canton, Ohio
  - Stark Pediatrics Inc., Canton, Ohio
  - Anderson Hills Pediatrics, Inc., Cincinnati, Ohio
  - Pediatric Associates of Mt. Carmel, Cincinnati, Ohio
  - Pediatric Associates of Fairfield, Fairfield, Ohio
  - Landen Lake Pediatrics, Mason, Ohio
  - Euclid Pediatrics, Mentor, Ohio
  - ESD Pediatric Group, Milford, Ohio
  - Crown Point Pediatrics, Toledo, Ohio
  - Pediatric Associates of Youngstown, Youngstown, Ohio
  - Pediatric Associates of Gresham, Gresham, Oregon
  - PMC, McMinnville, Oregon
  - Johnson Pediatrics, Medford, Oregon
  - Jo Anne Nielsen, MD, Oregon City, Oregon
  - Bellevue Pediatrics, Bellevue, Pennsylvania
  - PMA Medical Specialists, LLC, Collegeville, Pennsylvania
  - Franklin Street Pediatrics, Johnstown, Pennsylvania
  - Eden Park Pediatric, Lancaster, Pennsylvania
  - Praful Bhatt, MD, Lock Haven, Pennsylvania
  - Pediatrics South- Robinson, McKees Rock, Pennsylvania
  - McMurray Pediatric & Adolescent Medicine, McMurray, Pennsylvania
  - Red Lion Pediatrics, Philadelphia, Pennsylvania
  - Mt. Airy Pediatrics, LLP, Philadelphia, Pennsylvania
  - Cevallos & Moise Pediatrics, Quakertown, Pennsylvania
  - Pennridge Pediatric Associates, Sellersville, Pennsylvania
  - Susquehanna Int. Med. Pediatrics, Williamsport, Pennsylvania
  - Lake Area Pediatrics, Providence, Rhode Island
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Palmetto Medical Research, LLC, Mt. Pleasant, South Carolina
  - Plateau Pediatrics, Crossville, Tennessee
  - Siskiyou Pediatric Clinic, LLP, Crossville, Tennessee
  - Cool Springs Pediatrics, Franklin, Tennessee
  - Cumberland Pediatric Associates, Lebanon, Tennessee
  - Cedar Creek Pediatrics & Adolescent Medicine, Maryville, Tennessee
  - Sheffield Pediatrics, Memphis, Tennessee
  - Soddy Daisy Pediatrics, Soddy-Daisy, Tennessee
  - Pediatric Clinical Trials, LLC, Tullahoma, Tennessee
  - Jorge A Patino MD PA, Brownsville, Texas
  - Coppell Pediatrics, Coppell, Texas
  - Sarah L. Helfand, M.D., Dallas, Texas
  - Healthy Texan Pediatrics and Family Medicine, Dallas, Texas
  - Iresh Kumar MD, Frisco, Texas
  - Texas Childrens Pediatric Associates, Houston, Texas
  - Pediatric Associates, Houston, Texas
  - VIP Pediatrics, Houston, Texas
  - Pediatric Associates of Lubbock, Lubbock, Texas
  - Pediatric Care Associates, LLC, Montgomery, Texas
  - The Pediatric Clinic, P.A., Mount Pleasant, Texas
  - Pediatric Associates of North Texas, Plano, Texas
  - ChildCare Associates, San Antonio, Texas
  - Southwest Children's Research Associates, P.A., San Antonio, Texas
  - Tejas Pediatrics, Tejas, Texas
  - A Brighter Tomorrow Pediatrics, Webster, Texas
  - Sunshine Kids Medical Associates, Webster, Texas
  - Jean Brown Research-Odgen Clinic, Odgen, Utah
  - Utah Valley Pediatrics, Orem, Utah
  - Valle Verde Pediatrics, West Jordan, Utah
  - Van Dorn Pediatrics, Alexandria, Virginia
  - King George Pediatrics, King George, Virginia
  - Woodlake Village Pediatrics, Midlothian, Virginia
  - Richmond Pediatric Associates, Richmond, Virginia
  - Stafford Pediatrics, P.C., Stafford, Virginia
  - Redmond Pediatrics, Redmond, Washington
  - Elizabeth A. Tomeo, MD, Spokane, Washington
  - Community Pediatrics, Beaver Dam, Wisconsin
  - Pro Health Care Medical Associates, Muskego, Wisconsin
  - Lake Country Pediatrics, Oconomowoc, Wisconsin

REFERENCES:
- [Result] Toback SL, Carr W, Hackell J, Bhatt P, Ryan A, Ambrose CS. Influenza vaccination of parents and guardians by US pediatricians. Hum Vaccin. 2011 Apr;7(4):436-40. doi: 10.4161/hv.7.4.14171. Epub 2011 Apr 1. PMID 21445003
- [Result] Bhatt P, Block SL, Toback SL, Ambrose CS. Timing of the availability and administration of influenza vaccine through the vaccines for children program. Pediatr Infect Dis J. 2011 Feb;30(2):100-6. doi: 10.1097/INF.0b013e3181efff54. PMID 20686436
- [Result] Bhatt P, Block SL, Toback SL, Ambrose CS. A prospective observational study of US in-office pediatric influenza vaccination during the 2007 to 2009 influenza seasons: use and factors associated with increased vaccination rates. Clin Pediatr (Phila). 2010 Oct;49(10):954-63. doi: 10.1177/0009922810370868. Epub 2010 Jun 3. PMID 20522609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study of 118 physician offices in the USA identified the number of patients per practice by age group. A baseline survey and semi-monthly surveys of number of influenza vaccination doses given, staff attitudes toward influenza vaccination, and activities to increase influenza vaccination coverage were completed.
Pre-assignment Details: While a total of 147494 children were vaccinated in participating physicians' offices, no subjects were actually treated in this observational study.
Groups:
- Participants 9 to 18 Years: Pediatric influenza vaccine coverage within practicing pediatricians' offices for participants 9 to 17 years of age
Period: Overall Study
Arm/Group | Participants 6 to 23 Months | Participants 24 to 59 Months | Participants 5 to 8 Years | Participants 9 to 18 Years
Started | 28101 | 35967 | 36496 | 46930
Completed | 28101 | 35967 | 36496 | 46930
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants 6 to 23 Months | Participants 24 to 59 Months | Participants 5 to 8 Years | Participants 9 to 18 Years | Total
Number analyzed (Participants) | 28101 | 35967 | 36496 | 46930 | 147494
Age, Customized [Number; unit: participants] — Number of participants in each age group
  participants | 28101 | 35967 | 36496 | 46930 | 147494
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was not collected.
  Participants
    Female | NA — Gender was not collected. | NA — Gender was not collected. | NA — Gender was not collected. | NA — Gender was not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Gender was not collected. | NA — Gender was not collected. | NA — Gender was not collected. | NA — Gender was not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Influenza Vaccine Coverage in Participants <18 Years of Age by Age Group in Pediatric Practices
Description: Vaccine coverage was calculated from the number of participants vaccinated in each group, divided by the total number of participants under the practice's care in that specific age group.
Time Frame: Seasonal: 2007-2011
Measure: Number; unit: percentage of participants
Arm/Group | Participants 6 to 23 Months | Participants 24 to 59 Months | Participants 5 to 8 Years | Participants 9 to 18 Years
Number analyzed (Participants) | 28101 | 35967 | 36496 | 46930
percentage of participants | 46.5 | 30.9 | 30.6 | 19.4

2. Secondary Outcome: Compliance With the Recommended Two-dose Regimen in Vaccinated Participants
Description: Compliance was calculated from the total number of participants receiving 2 doses divided by the total number of participants identified as requiring a second dose.
Time Frame: Seasonal: 2007-2011
Measure: Number; unit: percentage of participants
Arm/Group | Participants 6 to 23 Months | Participants 24 to 59 Months | Participants 5 to 8 Years | Participants 9 to 18 Years
Number analyzed (Participants) | 28101 | 35967 | 36496 | 46930
percentage of participants | 67.5 | 42.7 | 40.8 | NA — Compliance was not calculated for this age group as 2 doses are not required.

3. Secondary Outcome: Correlation of Office Vaccination-related Attitudes and Activities With Actual Vaccine Coverage
Description: Correlation of office attitudes related to influenza vaccination and actual vaccine coverage was explored. Sites were asked to indicate level of agreement with the following recommendations: vaccinating children with high-risk medical conditions, patients 6 months to 5 years of age should be vaccinated against influenza each year, patients 5 to 18 years of age without high-risk medical conditions should be vaccinated against influenza each year, and previously unvaccinated patients less than 9 years of age receive 2 doses of vaccine.
Time Frame: Seasonal: 2007-2011
Measure: Number; unit: Sites
Groups:
- Staff Attitudes: High-risk Medical Conditions: Number of sites that agreed or somewhat agreed that they strongly recommend seasonal influenza vaccination to patients 5 to 18 years of age with high-risk medical conditions
- Staff Attitudes: 6 Months to 5 Year Old Patients: Number of sites that strongly recommend that patients 6 months to 5 years of age be vaccinated against influenza each year.
- Staff Attitudes: 5 to 18 Year Old Patients: Number of sites that agreed or somewhat agreed that they strongly recommend that patients 5 to 18 years of age without high-risk medical conditions be vaccinated against influenza each year
- Staff Attitudes: Number of Doses: Number of sites that agreed or somewhat agreed that they strongly recommend that previously unvaccinated patients less than 9 years of age receive 2 doses of influenza vaccine
Arm/Group | Staff Attitudes: High-risk Medical Conditions | Staff Attitudes: 6 Months to 5 Year Old Patients | Staff Attitudes: 5 to 18 Year Old Patients | Staff Attitudes: Number of Doses
Number analyzed (Participants) | 118 | 118 | 118 | 118
Sites | 117 | 118 | 118 | 117

ADVERSE EVENTS:
Groups:
- Children 6 to 23 Months; Children 24 to 59 Months; Children 5 to 8 Years; Children 9 to 18 Years: AEs were not collected in this observational study of physician vaccination practices.
Arm/Group | Children 6 to 23 Months | Children 24 to 59 Months | Children 5 to 8 Years | Children 9 to 18 Years
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.